CLINICAL TRIAL: NCT03596437
Title: Study of Arterial Properties by Ultra-high Frequency Ultrasound in Fibromuscular Dysplasia and Vascular Ehlers-Danlos Syndrome
Acronym: FUCHSIA-FR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P180201J
Record Dates: First submitted 2018-05-29; First posted 2018-07-23 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Ehlers-Danlos Syndrome; Fibromuscular Dysplasia
Keywords: Fibromuscular dysplasia; Vascular Ehler-Danlos Syndrome; Ultrasound
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Fibromuscular Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ehlers-Danlos Syndrome (Experimental): Intima-media thickness by ultrahigh frequency vs standard ultrasound
  Interventions: Device: Ultra High Frequency ultrasound system
- Fibromuscular Dysplasia (Experimental): Triple signal by ultrahigh frequency vs standard ultrasound
  Interventions: Device: Ultra High Frequency ultrasound system

INTERVENTIONS:
Device: Ultra High Frequency ultrasound system — Agreement for carotid intima-media thickness in vascular Ehlers Danlos Syndrome and for triple signal identification in fibromuscular dysplasia will be assessed.
  Other Names: Vevo MD

SUMMARY:
Ultra-high frequency ultrasound may be useful in the field of vascular research, given its ability to accurately characterize arterial wall thickness and ultrastructure.

In patients with fibromuscular dysplasia (FMD), it may help identify the "triple signal" pattern in carotid arterial wall, while in Vascular Ehlers Danlos Syndrome (V-EDS) it may help to accurately measure carotid intima-media thickness, which may be extremely small and difficult to measure with standard equipment. Furthermore, novel features might be identified in small-to-medium sized arteries by ultra-high frequency ultrasound.

The main aim of this study is to demonstrate that ultra-high frequency ultrasound has the same accuracy of standard ultrasound for the identification of "triple signal" in the carotid artery of FMD.

Secondary aims of this study are to evaluate carotid, radial and digital intima-media thickness, wall ultrastructure and distensibility in 60 patients with FMD and in 30 patients with V-EDS.

DETAILED DESCRIPTION:
Background: Fibromuscular dysplasia (FMD) is an idiopathic, systemic, non-atherosclerotic, non-inflammatory vascular disease leading to stenosis, aneurysms, dissections and occlusion of small and medium-sized arteries, with possible life-threatening complications. Recent data suggest that FMD is not so rare as previously thought, showing a prevalence up to 4%, but it is mostly undiagnosed. FMD mainly involves renal and internal carotid arteries, thus its clinical manifestations include hypertension and stroke. However, increasing evidence from large registries point out that FMD is a systemic disease, with a very high prevalence of multiple districts involvement.

Vascular Ehlers Danlos Syndrome (V-EDS) is a rare vascular disease (prevalence 1/150000), due to heterozygous mutations of COL3A1 gene, coding for collagen tipe III, with dominant autosomic transmission. V-EDS patients are predisposed to spontaneous ruptures in the vascular, intestinal districts and in many others.

In FMD, vascular subclinical alterations may be observed in usually usually not affected arterial districts, such as the common carotid artery and the radial artery. In a previous experience, Boutouyrie and colleagues discovered a peculiar phenotype in the common carotid artery of individuals with renal FMD. This pattern, known as "triple signal", is characterized by a supernumerary acoustic interface, located between the blood-intima and the media- adventitia interfaces and detected by either the B-mode or the radiofrequency equipment, which may correspond to medial hyperplasia. The "triple signal" pattern, though present in a small proportion of hypertensive patients, was able to accurately discriminate FMD individuals and in particular to identify familiar cases. Furthermore, c-IMT was higher in FMD, while diameter and elasticity were superimposable to hypertensive control group.

Nevertheless, the study of non-affected and easily accessible medium and small-sized arteries, such as the radial artery, with similar diameter and histology of affected arteries such as the renal, cerebral and coronary arteries, might be even more informative in FMD. This has been recently made possible by the commercial availability of ultra-high frequency ultrasound for human use. The machine is equipped with transducers up to 70 MHz and allows imaging superficial tissues with a spatial resolution up to 30 μm (axial) and 65 μm (lateral). Preliminary results by using ultrahigh frequency ultrasound, confirmed an increased radial wall thickness in FMD patients in comparison to age-, sex- and BP-matched controls. Most strikingly, wall ultrastructure was extensively subverted in FMD patients: the two echogenic layers corresponding to the elastic laminae presented a lower echogenicity and a greater inhomogeneity as compared to healthy individuals.

Methods: This is a cross-sectional study, recruiting 60 individuals with FMD and 30 individuals with V-EDS. Patients will be recruited by the Clinical Pharmacology Unit of the Hopital Europeen George Pompidou, during their routine visit for the ultrasound evaluation of the carotid arteries by echotracking. In that occasion, supplementary images of carotid, radial and digital arteries will be acquired by ultrahigh frequency ultrasound (VevoMD; Fujifilm-Visualsonics: Toronto, Canada).

ELIGIBILITY:
Inclusion Criteria for patients with FMD:

* Patients aged between 18 and 80 inclusive
* Patients who have already been diagnosed with FMD of the renal arteries, cervical or cerebral arteries or spontaneous coronary dissections
* Informed consent signed,
* Patient affiliated to a social security.

Inclusion Criteria for patients with Ehlers-Danlos vascular syndrome:

* Patients aged between 18 and 80 inclusive
* Patients with a previous diagnosis of vascular Ehlers-Danlos vascular syndrome
* Informed consent signed,
* Patient affiliated to a social security.

Exclusion Criteria:

* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the Public Health Code
* Person subject to an exclusion period for another research
* Pregnancy in progress
* Allergies to ultrasound gel or skin lesions (severe eczema, wounds, etc.) that prevent the echo probe from being applied to the area of interest.
* Refusal or inability to read information, to sign informed consent and not to oppose research, linguistically or psychologically
* Severe life-threatening disease in the short to medium term

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Agreement between ultrahigh-frequency and standard ultrasound in the identification of "triple signal" in the common carotid artery wall in fibromuscular dysplasia | through study completion (an average of 30 minutes)
  Triple signal is defined as the visual identification of supernumerary acoustic interface in the common carotid artery wall; K statistics will be used.

SECONDARY OUTCOMES:
Agreement between ultrahigh frequency and standard ultrasound in the evaluation of carotid intima-media thickness in fibromuscular dysplasia. | through study completion (an average of 30 minutes)
Agreement between ultrahigh frequency and standard ultrasound in the evaluation of carotid intima-media thickness in vascular Ehlers-Danlos syndrome. | through study completion (an average of 30 minutes)
Agreement between ultrahigh frequency and standard ultrasound in the evaluation of carotid distensibility in fibromuscular dysplasia. | through study completion (an average of 30 minutes)
Agreement between ultrahigh frequency and standard ultrasound in the evaluation of carotid distensibility in vascular Ehlers-Danlos syndrome. | through study completion (an average of 30 minutes)
Reproducibility of radial intima-media thickness, measured by ultrahigh frequency ultrasound in fibromuscular dysplasia and vascular Ehlers-Danlos syndrome. | through study completion (an average of 30 minutes)
  Intraclass coefficient, correlation at will be used
Reproducibility of radial distensibility, measured by ultrahigh frequency ultrasound in fibromuscular dysplasia and vascular Ehlers-Danlos syndrome. | through study completion (an average of 30 minutes)
  Intraclass coefficient, correlation at will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de pharmacologie clinique HEGP, Paris, France

IPD SHARING:
Plan to Share IPD: No